CLINICAL TRIAL: NCT02840188
Title: Young Goalkeeper's Fracture: Radiographic Findings, Risk Factors and Prevention Measures
Brief Title: Young Goalkeeper's Fracture: Radiographic Findings
Acronym: Goalkeeper
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-BE: 2016-00670
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Radius Fractures
Keywords: goalkeeper's fracture
MeSH Terms: conditions — Radius Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Radius tilt angle: Children 0-16 years of age positive for distal forearm fracture and positive history of goalkeeper's fracture (to catch a ball).
  Interventions: Other: Radius tilt angle
- Normal control group: Children 0-16 years of age without radius fracture and no history of catching a ball.
  Interventions: Other: Radius tilt angle

INTERVENTIONS:
Other: Radius tilt angle — Fracture classification in children. Tilt angle measurement of the distal radius growth plate.

SUMMARY:
The aim of this project is to evaluate retrospectively goalkeeper's fractures in children using the children fracture classification and to evaluate the distal radius tilt angle of the growth plate on plain radiographs of the forearm.

Patients positive for goalkeeper's fracture will prospectively answer a questionnaire concerning risk factors and circumstances during the injury.

DETAILED DESCRIPTION:
Distal forearm or radius fractures in young goalkeepers have been named "the young goalkeeper's fracture" in the literature. While catching the soccer ball the child suffers a distal forearm fracture due to axial forces to the immature bone of the child. These goalkeeper's fractures on radiographs may be subtle or difficult to discriminate from normal radiographs.

Retrospective study for the evaluation of radiographs of the forearm from 2005 - 2016 of children with history of catching a ball. Two radiologist are blinded for history, age, name and findings on final reports.

First reading without measurement of distal tilt angle, second reading with measurement of distal tilt angle and after consensus meeting.

Questionnaire: prospectively all patients with goalkeeper's fracture will answer a questionnaire concerning circumstances and risks during the accident.

ELIGIBILITY:
Inclusion Criteria:

* Children 1-16 years of age with distal radius fracture and the clinical history: "child catches a ball", between 1/2005 - 7/2016.
* Control group (1-16 years) with normal distal radius and no history to catch a ball and no fracture.

Evaluation of the normal distal tilt angle of the radius.

Exclusion Criteria:

* pathological fractures
* other history of trauma than to catch a ball
* patients older than 16 years

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Distal radius fracture in young goalkeepers (=young goalkeeper's fracture)
Sampling Method: Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Tilt angle of distal radius growth plate in goalkeeper's fracture | 2005- 2016
  Dorsal angulation of distal radius growth plate in goalkeeper's fracture

SECONDARY OUTCOMES:
Risk factors for goalkeeper's fracture | 2005-2016
  Questionnaire for circumstances and risks for goalkeeper's fracture

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Heverhagen, MD, Study Chair — University Hospital Bern, Inselspital
Locations (1):
- University Hospital Berne, Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boyd KT, Brownson P, Hunter JB. Distal radial fractures in young goalkeepers: a case for an appropriately sized soccer ball. Br J Sports Med. 2001 Dec;35(6):409-11. doi: 10.1136/bjsm.35.6.409. PMID 11726476
- [Background] Kraus R, Szalay G, Meyer C, Kilian O, Schnettler R. [Distal radius fracture - a goalkeepers' injury in children and adolescents]. Sportverletz Sportschaden. 2007 Dec;21(4):177-9. doi: 10.1055/s-2007-963706. German. PMID 18072076